CLINICAL TRIAL: NCT06939335
Title: The Application of Positive End-Expiratory Pressure in Out-of-Hospital Cardiac Arrest: The Lazarus-PEEP Trial.
Acronym: Lazarus-PEEP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ONZ-2024-0496
Record Dates: First submitted 2025-03-31; First posted 2025-04-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Arrest (CA); Out-of-hospital Cardiac Arrest (OHCA); Positive End-expiratory Pressure (PEEP); Ventilation During Resuscitation
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Intervention Model Description: Multicenter parallel controlled randomised clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Ventilation during cardiac arrest with an adult Resuscitation Bag with a pressure relief valve set at 40 cm H20 and a disposable PEEP Valve set at 5 cm H20.
  Interventions: Device: Disposable PEEP Valve set at 5 cm H20.
- Controle (Active Comparator): Ventilation during cardiac arrest with an adult Resuscitation Bag with a pressure relief valve set at 40 cm H20 without a disposable PEEP Valve.
  Interventions: Device: Controle

INTERVENTIONS:
Device: Disposable PEEP Valve set at 5 cm H20. — Ventilation during cardiac arrest with an adult Resuscitation Bag with a pressure relief valve set at 40 cm H20 and a 22 mm disposable PEEP Valve set at 5 cm H20.
  Arms: Intervention
Device: Controle — Ventilation during cardiac arrest with an adult Resuscitation Bag with a pressure relief valve set at 40 cm H20 without a disposable PEEP Valve.
  Arms: Controle

SUMMARY:
The goal of this clinical trial is to learn whether using Positive End-Expiratory Pressure (PEEP) during cardiopulmonary resuscitation (CPR) improves outcomes for adults who experience out-of-hospital cardiac arrest, a condition where the heart suddenly stops beating. PEEP is used during ventilation, which may enhance oxygen levels by keeping the airways open throughout CPR.

This study aims to determine if using PEEP during CPR helps restart the heart more effectively, improves survival rates, and enhances survival with good neurologic outcomes after a cardiac arrest compared to standard CPR without PEEP.

Researchers will randomly assign participants to one of two groups: one receiving CPR with PEEP set at 5 cm of water pressure and the other receiving standard CPR without PEEP. Participants will be treated by emergency medical teams trained in advanced life support, and specialised sensors will measure airflow and airway pressure during resuscitation.

Additionally, the study will evaluate potential side effects associated with PEEP, such as increased pressure within the chest or lung injuries. Findings from this trial will guide recommendations on the usage of PEEP in standard CPR practices to potentially improve patient outcomes.

DETAILED DESCRIPTION:
Introduction: Sudden cardiac arrest is a significant cause of mortality, with an estimated annual incidence of 84 cases per 100,000 individuals in Europe. Effective cardiopulmonary resuscitation (CPR), including proper ventilation, is crucial for survival. However, the interplay between ventilation and circulation during CPR is complex and not fully understood. While ventilation is necessary for oxygenation, excessive hyperventilation and high intrathoracic pressures can be detrimental. Positive End-Expiratory Pressure (PEEP) may improve oxygenation and ventilation by maintaining alveolar patency and improving oxygenation. Previous observational studies have suggested that PEEP might enhance the rate of Return of Spontaneous Circulation (ROSC) and improve short-term outcomes. However, no prospective randomised clinical trials have been conducted to confirm these findings. The Lazarus-PEEP trial aims to address this gap by evaluating the efficacy and safety of PEEP during CPR for out-of-hospital cardiac arrest (OHCA) patients.

Methodology: The study will be conducted at Ghent University Hospital and three non-university hospitals in Belgium, enrolling adult patients who experience non-traumatic OHCA and are intubated and ventilated during resuscitation efforts by an advanced life support (MUG) team. Participants will be randomised to receive either PEEP at 5 cm H2O or no PEEP (0 cm H2O) during CPR. Custom-built sensors will measure tracheal airflow and pressure, while additional data on CPR quality and patient outcomes will be collected. The trial's primary outcome measure is the rate of ROSC, with secondary outcomes including survival to hospital admission and discharge, as well as neurological outcomes at discharge.

Outcome: The study will evaluate the effectiveness of PEEP in improving ROSC rates, short-term survival, and neurological outcomes. Safety profiles will also be examined, focusing on adverse effects such as barotrauma and increased intrathoracic pressures. Comprehensive data collection will provide insights into the physiological impact of PEEP during CPR and its feasibility in a pre-hospital setting.

Conclusion: The Lazarus-PEEP trial aims to gather strong evidence on the potential advantages and risks of utilizing PEEP during CPR for OHCA patients. The results will inform evidence-based guidelines and enhance resuscitation practices, potentially leading to improved patient outcomes. The findings will be disseminated through influential journals, major scientific conferences, and public data-sharing platforms to ensure widespread accessibility and impact.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Adults aged 18 years and older.
2. Type of Cardiac Arrest: Patients who have experienced a non-traumatic out-of-hospital cardiac arrest.
3. CPR Administration: Patients receiving cardiopulmonary resuscitation from an advanced life support (ALS) team.
4. Intubation and Ventilation: Patients who are intubated and ventilated during resuscitation efforts.

Exclusion Criteria:

1. Cardiac arrest in patient younger than 18 years of age.
2. Traumatic cardiac arrest, including drowning, penetrating or blunt injury, and burns.
3. Immediate Return of Spontaneous Circulation (ROSC): Patients who achieve ROSC before intubation and initiation of intubation.
4. Pregnancy.
5. Mechanical ventilation during arrest: patients already receiving mechanical ventilation at the moment of cardiac arrest, due to reasons other than their arrest, will be excluded.
6. Do Not Resuscitate (DNR) Orders: Patients with existing DNR orders or any advanced directive indicating that CPR should not be performed.
7. Failure to intubate: if intubation is unsuccessful, ventilation by any means (MBV, SGA) should take priority over the study protocol, and the patient is excluded.
8. Enrolment in Other Studies: Patients currently enrolled in another interventional clinical trial that could interfere with the outcomes of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Return of spontaneous circulation (ROSC) | Day one
  The occurrence of Return of spontaneous circulation (ROSC), defined as the return of sustained spontaneous circulation for at least 20 minutes per ERC guidelines

SECONDARY OUTCOMES:
Survival to hospital admission | Day one
Survival to hospital discharge | From enrolment until hospital discharge or death - whichever happens first. Average hospitalisation after OHCA is 24 days.
30-day survival | From enrollment to the end of 30 days.
90-day survival | From enrollment to the end of 90 days.
Neurological outcome at discharge | From enrolment until hospital discharge or death - whichever happens first. Average hospitalisation after OHCA is 24 days.
  Neurological outcome at discharge, as defined by the Cerebral Performance Category Scale.

OTHER OUTCOMES:
Airflow during ventilation | Periprocedural
  The Sensirion SFM3200AW flow sensor will measure airflow during cardiopulmonary resuscitation, measured in ml.
Airway pressure during ventilation | Periprocedural
  The Wika CPT2500 sensor will measure airway pressure during cardiopulmonary resuscitation, measured in mbar.
Occurence of potential adverse effects | Day one
  The incidence of barotrauma, including pneumothorax and pneumomediastinum
Capnography | Periprocedural
  the ZOLL® X Series® monitor-defibrillator will be used to collect capnography data during cardiopulmonary resuscitation, measured in mmHg.
Compression depth | Periprocedural
  The ZOLL® X Series® monitor-defibrillator will be used to measure Compression depth, measured in mm.
Compression frequency | Periprocedural
  The ZOLL® X Series® monitor-defibrillator will be used to measure Compression frequency, measured in compressions/minute.

CONTACTS AND LOCATIONS:
Overall Officials: Saïd Hachimi Idrissi, MD, PhD, Professor, Principal Investigator — UZ Gent
Locations (7):
- Belgium (6):
  - AZ Oostende, Ostend, West-Flandres
  - AZORG: campus Merestraat, Aalst
  - AZORG: Campus Moorselbaan, Aalst
  - AZORG: campus Geraardsbergen, Geraardsbergen
  - UZ Ghent, Ghent
  - AZ Zeno, Knokke
- Centre hospitalier universitaire (CHU) Besançon-Franche-Comté, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided